CLINICAL TRIAL: NCT02190942
Title: VCRC Validation of Patient-Reported Diagnostic Data
Brief Title: VCRC Patient Contact Registry Patient-Reported Data Validation Study
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Wayne State University (Other); University of Pittsburgh (Other); University of Pennsylvania (Other); Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: 5535
Record Dates: First submitted 2014-05-30; First posted 2014-07-15 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Behcet's Disease; Churg-Strauss Syndrome; Giant Cell Arteritis; Wegener Granulomatosis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu's Arteritis
MeSH Terms: conditions — Behcet Syndrome; Churg-Strauss Syndrome; Giant Cell Arteritis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vasculitis Contact Registry Patients: Consent will be obtained from at least 20 randomly selected patients with each of the following self-identified diagnoses in the VCRC Patient Contact Registry: Behçet's disease, EGPA, GCA, GPA, MPA, PAN and TAK that have already completed the VCRC Diagnostic Questionnaires. Permission will be obtained to contact subjects' primary vasculitis care providers to request that the providers complete an online version of this questionnaire (or print copy, if they prefer), and request specific chart items from their office to further verify the data.

SUMMARY:
The purpose of this study is to provide validation of patient-reported data in the VCRC Patient Contact Registry by comparing patient-reported data with data provided by the physician who is the primary provider caring for the patient's vasculitis. Patients enrolled in the Patient Contact Registry with Behcet's disease, eosinophilic granulomatosis with polyangiitis (Churg-Strauss) (EGPA), giant cell arteritis (GCA), granulomatosis with polyangiitis (Wegener's) (GPA), microscopic polyangiitis (MPA), polyarteritis nodosa (PAN), and Takayasu's arteritis (TAK) were invited via email to participate in this study.

DETAILED DESCRIPTION:
Via email, consent was obtained from at least 20 randomly selected patients with the seven forms of vasculitis detailed above in the VCRC Patient Contact Registry who have completed the Diagnostic Questionnaire. The form was sent in PDF format to the patient, who either printed out or emailed the form to his or her primary vasculitis provider to complete. This form included the same questions in the patient questionnaire, with minor reformatting and a few expanded details to verify the patient-provided data (please see appendix B). If the 20 questionnaires are not returned one month after the initial recruitment email to the Patient Contact Registry participants, 20 additional participants with the seven forms of vasculitis will be selected randomly and will be asked to participate in this study. The survey data is stored by the Rare Diseases Clinical Research Network's (RDCRN) Data Management and Coordinating Center (DMCC) at the University of South Florida. The data is de-identified. Names or other personal health information were not collected. Upon conclusion of the study period, the data will be sent to Dr. Kathleen McKinnon. All data collected will be sent to the database of Genotypes and Phenotypes (dbGaP) to be stored indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 patients with each of the following self-identified diagnoses in the VCRC Patient Contact Registry: Behçet's disease, EGPA, GCA, GPA, MPA, PAN, and TAK who have completed the online questionnaires.

Exclusion Criteria:

* Inability to provide informed consent and complete survey
* Patients whose diagnosis of vasculitis was not confirmed by a physician
* Patients who did not complete the initial questionnaire in its entirety

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consent will be obtained from at least 20 randomly selected patients with each of the following self-identified diagnoses in the VCRC Patient Contact Registry: Behçet's disease, EGPA, GCA, GPA, MPA, PAN and TAK that have already completed the VCRC Diagnostic Questionnaires. Permission will be obtained to contact subjects' primary vasculitis care providers to request that the providers complete an online version of this questionnaire (or print copy, if they prefer), and request specific chart items from their office to further verify the data. The sensitivity and specificity for various combinations of the diagnostic questions to predict vasculitis and to confirm type of vasculitis will be calculated using physician diagnosis / chart review as the gold standard.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Validation of the currently utilized VCRC Patient Contact Registry Questionnaire | Up to 24 months from the date of the last patient assessment
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

SECONDARY OUTCOMES:
Evaluate diagnostic accuracy of specific questions | Up to 24 months form the last patient assessment received
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen McKinnon, DO, Study Chair — Henry Ford/Wayne State University; Ximena D. Ruiz, MD, Study Chair — University of Pittsburgh; Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania; Jennifer L. Harris, MSPH, CCRP, Study Chair — University of South Florida
Locations (1):
- University of South Florida Data Management Coordinating Center, Tampa, Florida, United States